CLINICAL TRIAL: NCT05172258
Title: A Phase 2 Study of Ipatasertib in Combination With Pembrolizumab for First Line Treatment of Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck
Brief Title: Testing the Addition of an Anti-cancer Drug, Ipatasertib, to the Usual Immunotherapy Treatment (Pembrolizumab) in Patients With Recurrent or Metastatic Squamous Cell Cancer of the Head and Neck
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-13902; NCI-2021-13902 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PHII-216; 10496 (Other: City of Hope Comprehensive Cancer Center LAO); 10496 (Other: CTEP); UM1CA186717 (NIH)
Record Dates: First submitted 2021-12-28; First posted 2021-12-29 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma; Metastatic Hypopharyngeal Squamous Cell Carcinoma; Metastatic Laryngeal Squamous Cell Carcinoma; Metastatic Oral Cavity Squamous Cell Carcinoma; Metastatic Oropharyngeal Squamous Cell Carcinoma; Recurrent Head and Neck Squamous Cell Carcinoma; Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Oral Cavity Squamous Cell Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Stage IV Hypopharyngeal Carcinoma AJCC v8; Stage IV Laryngeal Cancer AJCC v8; Stage IV Lip and Oral Cavity Cancer AJCC v8; Stage IV Oropharyngeal (p16-Negative) Carcinoma AJCC v8
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Carcinoma | interventions — Biopsy; Specimen Handling; ipatasertib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (ipatasertib, pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 and ipatasertib PO QD on days 1-14 of each cycle. Cycles repeat every 21 days for a period of 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, undergo collection of blood samples on study and during follow up, and undergo CT scans throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Drug: Ipatasertib; Biological: Pembrolizumab
- Arm II (pembrolizumab) (Active Comparator): Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for a period of 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, undergo collection of blood samples on study and during follow up, and undergo CT scans throughout the trial.
  Interventions: Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Biological: Pembrolizumab

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Ipatasertib — Given PO
  Other Names: GDC 0068; GDC-0068; GDC0068; RG 7440; RG-7440; RG7440
  Arms: Arm I (ipatasertib, pembrolizumab)
Biological: Pembrolizumab — Given IV
  Other Names: BCD-201; GME 751; GME751; Keytruda; Lambrolizumab; MK 3475; MK-3475; MK3475; Pembrolizumab Biosimilar BCD-201; Pembrolizumab Biosimilar GME751; Pembrolizumab Biosimilar QL2107; Pembrolizumab Biosimilar RPH-075; Pembrolizumab Biosimilar SB27; QL2107; RPH 075; RPH-075; RPH075; SB 27; SB-27; SB27; SCH 900475; SCH-900475; SCH900475

SUMMARY:
This phase II trial compares the effect of adding ipatasertib to pembrolizumab (standard immunotherapy) vs. pembrolizumab alone in treating patients with squamous cell cancer of the head and neck that has come back (recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Ipatasertib is in a class of medications called protein kinase B (AKT) inhibitors. It may stop the growth of tumor cells and may kill them. Immunotherapy with monoclonal antibodies, such as pembrolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving ipatasertib in combination with pembrolizumab may be more effective than pembrolizumab alone in improving some outcomes in patients with recurrent/metastatic squamous cell cancer of the head and neck.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare progression-free survival (PFS) in first line relapsed/metastatic (R/M) head and neck squamous cell cancer (HNSCC) patients treated with the combination ipatasertib and pembrolizumab versus pembrolizumab monotherapy treatment.

SECONDARY OBJECTIVES:

I. To evaluate the safety and tolerability of the combination ipatasertib and pembrolizumab in first line R/M HNSCC patients.

II. To describe overall response rate (ORR) and duration of response per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 in first line R/M HNSCC treated patients with the combination ipatasertib and pembrolizumab and pembrolizumab monotherapy treatment.

III. To assess changes in the tumor microenvironment by immunophenotyping with the combination ipatasertib and pembrolizumab and pembrolizumab monotherapy treatment.

IV. To assess changes in Akt, ERK, and MEK signaling with the combination ipatasertib and pembrolizumab and pembrolizumab monotherapy treatment.

V. To determine changes in immune-cell population in peripheral blood with the combination ipatasertib and pembrolizumab and pembrolizumab monotherapy treatment.

EXPLORATORY OBJECTIVE:

I. To investigate the relationship between the combination ipatasertib and pembrolizumab treatment and biomarkers which may predict response, such as tumor PD-L1 expression and alterations in the PI3K/AKT pathway.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 and ipatasertib orally (PO) once daily (QD) on days 1-14 of each cycle. Cycles repeat every 21 days for a period of 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, undergo collection of blood samples on study and during follow up, and undergo computed tomography (CT) scans throughout the trial.

ARM II: Patients receive pembrolizumab IV over 30 minutes on day 1 of each cycle. Cycles repeat every 21 days for a period of 24 months in the absence of disease progression or unacceptable toxicity. Patients also undergo biopsy on study, undergo collection of blood samples on study and during follow up, and undergo CT scans throughout the trial.

After completion of study treatment, patients are followed every 3 months until disease progression, the next line of therapy is started, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed recurrent or metastatic HNSCC that is considered incurable.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) by chest x-ray or as >=10 mm (>= 1 cm) with CT scan, magnetic resonance imaging (MRI), or calipers by clinical exam.
* Primary tumor locations of oral cavity, oropharynx, hypopharynx, and larynx are allowed. Participants may not have a primary tumor site of nasopharynx.
* Patients with oropharyngeal cancer must have known human papillomavirus (HPV) status defined by human papillomavirus type 16 (p16) testing.
* Patients should not have had prior systemic therapy administered in the recurrent or metastatic setting. Systemic therapy which was given as part of multimodal treatment for locally advanced disease is allowed.
* Patients must be able to provide an archival tissue specimen.
* Patients must be willing to undergo a mandatory tumor biopsy on treatment
* Tumor tissue must have a documented combined positive score (CPS) of >= 1 for PD-L1.
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of ipatasertib in combination with pembrolizumab in patients < 18 years of age, children are excluded from this study.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 (Karnofsky >= 60%).
* Absolute neutrophil count >= 1,000/mcL.
* Platelets >= 100,000/mcL.
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN).
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN.
* Creatinine =< 1.5 x institutional ULN.
* Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 (using the Cockcroft-Gault formula).
* Human immunodeficiency virus (HIV) infected patients on effective antiretroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Patients must be able to swallow orally administered medication whole.
* For women of childbearing potential (WOCBP): agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods with a failure rate of < 1% per year during the treatment period, for 5 months after the last dose of pembrolizumab and 28 days after the last dose of ipatasertib, and agreement to refrain from donating eggs during this same period.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, agreement to refrain from donating sperm during the treatment period, and for 5 months after the last dose of pembrolizumab and 28 days after the last dose of ipatasertib.
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) who have a legally-authorized representative (LAR) and/or family member available will also be eligible.

Exclusion Criteria:

* Prior treatment with a checkpoint inhibitor given for relapsed or metastatic disease. Prior treatment with a checkpoint inhibitor for locally advanced disease as part multidisciplinary treatment is allowed.
* History of malabsorption syndrome or other condition that would interfere with enteral absorption or result in the inability or unwillingness to swallow pills.
* Patient has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the study principal investigator (PI).
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine or physiologic corticosteroid replacement for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Type 1 or Type 2 diabetes mellitus requiring insulin at study entry are ineligible.

  * Patients who are on a stable dose of oral diabetes medication >= 4 weeks prior to initiation of study treatment may be eligible for enrollment. Patients must meet the laboratory eligibility criteria for fasting blood glucose and hemoglobin A1c.
  * Fasting glucose =< 150 mg/dL (8.3 mmol/L) and hemoglobin A1c =< 7.5% (58 mmol/mol).
* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1). Note: Patients with grade =< 2 neuropathy or grade =< 2 alopecia are an exception to this criterion and may qualify for the study. Note: If patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* Patients who are receiving any other investigational agents.
* Patients with known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ipatasertib or hypersensitivity (grade >= 3) to pembrolizumab and/or any of the components of the solution for injection.
* Treatment with strong CYP3A inhibitors or strong CYP3A inducers within 2 weeks or 5 drug-elimination half-lives, whichever is longer, prior to initiation of study drug is prohibited. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients with uncontrolled intercurrent illness (including but not limited to interstitial lung disease or active, non-infectious pneumonitis) or a history of (non-infectious) pneumonitis that required steroids.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Patients who are pregnant or breastfeeding, or are expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 5 months after the last dose of study treatment. A WOCBP who has a positive urine pregnancy test (e.g., within 72 hours) prior to treatment will be excluded from the study. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Pregnant women are excluded from this study because pembrolizumab is a monoclonal antibody agent and ipatasertib is an oral AKT inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pembrolizumab and ipatasertib, breastfeeding should be discontinued if the mother is treated with pembrolizumab or ipatasertib. Due to the potential risks, WOCBPs and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 5 months after the last dose of pembrolizumab and 28 days after the last dose of ipatasertib. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
* Patients with grade >= 2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia are excluded.
* Patient has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer) that has undergone potentially curative therapy.
* History of or active inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis).
* Lung disease: pneumonitis, interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia).
* Known clinically significant history of liver disease consistent with Child Pugh Class B or C, including active viral or other hepatitis (e.g., positive for hepatitis B surface antigen [HbsAg] or hepatitis C virus [HCV] antibody at screening), current drug or alcohol abuse, or cirrhosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until disease progression, death, or date of last contact, whichever occurs first, assessed up to 1 year after the last patient is enrolled
  The 1-sided log rank test for equality of risk for PFS-event will be performed (Dang et al., 2020). If the p-value is less than or equal to 0.15, it will be concluded that the ipatasertib plus pembrolizumab has sufficient efficacy for further evaluation.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 1 year after the last patient is enrolled
  Tables will be created to summarize the numbers of patients who experienced toxicities (graded according to the Common Terminology Criteria for Adverse Events version 5.0), by arm, toxicity system, type, grade, and attribution.
Overall response rate | Up to 1 year after the last patient is enrolled
  Will be assessed according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 for both cohorts in the study. The primary analysis will be based on a modified intention-to-treat analysis which will include all eligible, randomized patients who receive any amount of treatment according to the patient's randomization. The two arms will be compared in terms of the overall response rate (probability of complete response [CR] or partial response [PR] by RECIST version 1.1) using a one-sided, 0.10-level Mantel-Haenszel. Two-sided 80% confidence intervals will be constructed for the probability of response in each arm. In addition, a logistic regression (exact, if required based on the numbers) will be used to estimate the odds ratio comparing the 2 arms adjusting for the stratification variables.
Duration of response | From the date of the scan that first documented a PR or CR until the patient demonstrates a PFS event, assessed up to 1 year after the last patient is enrolled
  Will be assessed according to RECIST 1.1 for both cohorts in the study. Will be calculated as the date of the scan that first demonstrated a PR or CR until the patient demonstrates a PFS-event.
Changes in the tumor microenvironment by immunophenotyping | Baseline up to 1 year after the last patient is enrolled
  Will be assessed by comparing immunophenotype of paired biopsy specimens for individual patients, with archival/pre-treatment biopsy and the C2D7 biopsy. Categorical data methods, including exact conditional methods, will be used to compare the proportions of these various response categories across randomized treatment assignment.
Changes in Akt, ERK, and MEK signaling | Baseline up to 1 year after the last patient is enrolled
  Categorical data methods, including exact conditional methods, will be used to compare the proportions of these various response categories across randomized treatment assignment.
Changes in immune-cell population in peripheral blood | Baseline up to 1 year after the last patient is enrolled
  Will be assessed by comparing blood specimens for individual patients over time: baseline, defined as the blood sample obtained closest to but not exceeding the date of the first dose of protocol therapy; on day 7 of cycle 2; on day 1 of every odd cycle; and at progression while the patient is receiving combination therapy. The statistical null hypothesis is defined as no change in percent of each cell type across time points and between regimens. These will be assessed quantitatively using a non-parametric analysis of variance with time point and randomized regimen as predictor variables.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob S Thomas, Principal Investigator — City of Hope Comprehensive Cancer Center LAO
Locations (20):
- United States (20):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - City of Hope Antelope Valley, Lancaster, California
  - Keck Medicine of USC Koreatown, Los Angeles, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - USC Norris Oncology/Hematology-Newport Beach, Newport Beach, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - University of Texas Medical Branch, Galveston, Texas
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-04-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT05172258/ICF_000.pdf